CLINICAL TRIAL: NCT04392674
Title: Safety and Efficacy of Using the New Tissue Containment System With Hard Pipes Which Can Assemble With Detachable Trocars Seamlessly for Tissue Removal During Laparoscopic Myomectomy Morcellation
Brief Title: Safety and Efficacy of Using the New Tissue Containment System During Laparoscopic Myomectomy Morcellation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing Liang (Other)
Responsible Party: Sponsor-Investigator, Jing Liang, professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTCS-20200508
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gynecologic Surgery
Keywords: morcellation; myomectomy; laparoscopic surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- using the new tissue containment system (Experimental): using the new tissue containment system during Laparoscopic myomectomy morcellation
  Interventions: Device: the new tissue containment system

INTERVENTIONS:
Device: the new tissue containment system — using the new tissue containment system during Laparoscopic myomectomy morcellation

SUMMARY:
The study is designed to evaluate the safety of performing the new tissue containment system during laparoscopic myomectomy morcellation. Pre- and perimenopausal women, aged 18-45 undergoing laparoscopic myomectomy morcellation

ELIGIBILITY:
Inclusion Criteria:

* Pre- and Peri-menopausal woman patient age 18-45 years

  * Women with fibroids and indication for laparoscopic myomectomy.
  * Normal Pap smear result within one year
  * MRI ( Magnatic Resonance Imaging ) or other imaging findings indicate the diameter of the largest uterine fibroids is between 4 to 10cm.
  * The body mass index of the patients is 18.5-27.9kg/m2
  * Signed informed consent form

Exclusion Criteria:

* • Women with Known or suspected malignancy

  * patients with severe pelvic adhesion found during the operation
  * The body mass index of the patient ≥ 28kg/m2
  * Diameter of a single uterine fibroid>10cm
  * patients during pregnancy and lactation
  * Known blood diseases, bleeding coagulation disease, any part of the active bleeding or bleeding tendency of the constitution of the patient
  * Patients with known severe liver and kidney dysfunction;Liver function (ALT, AST) ≥ 2 times of normal upper limit, or renal function (Cr) ≥ normal upper limit
  * Patients who are known to have participated in any other clinical trial within 3 months
  * Patients who cannot sign informed consent
  * Patients with acute stage infection of the reproductive system or other sites

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
The safety of using the new tissue containment system for contained cutting and extracting tissue during laparoscopic myomectomy morcellation | approximately two years
  The safety of using the new tissue containment system for cutting and extracting tissue during laparoscopic myomectomy morcellation will be determined by the rate of leakage
  Leakage is defined as "disruption of the device (using dye leak testing) or visible tissue dissemination.

SECONDARY OUTCOMES:
The probability of failure during in-bag morcellation procedure | approximately two years
  Failure is defined as the operator's inability to successfully insert and extract the device.
Mean procedure time | approximately two years
  Mean procedure time will be measured by hour/minutes.
Estimated blood loss during operation | approximately two years
  Blood loss during operation will be measured by volume (mL)
Post-operative pain | approximately two years
  Post-operative pain will be measured by Visual Analog Score - VAS
Intra- or post-operative complications | approximately two years
  Intra or post complications rate (e.g. urinary, intestinal or nerve injury)
The Surgeon Task Load Index | approximately two years
  The Surgeon Task Load Index be measured by designated Questionnaire.
The Patients' life quality postoperative | approximately two years
  The Patients' life quality postoperative be measured by Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will to be shared with other researchers after four years